## SAPPHIRE II PRO Protocol Number: VP-0714 16 Feb 2017, Clinical Protocol V 1.0



# Statistical Analysis Plan

Protocol number: VP-0714rev 1.0

The **SAPPHIRE II PRO** Study

#### Confidential Information

The information contained in this Statistical Analysis Plan (SAP) is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Mount Sinai Heart or its subsidiaries. This document and its associated attachments or appendices are subject to United States Freedom of Information Act Exemption 4.

| TRIAL FULL TITLE | SAPPHIRE II PRO Study |
|---|---|
| PROTOCOL NUMBER | VP-0714 |
| SAP VERSION | 1.0 |
| SAP VERSION DATE | 25 September 2017 |
| SPONSOR | OrbusNeich, Medical, Inc. |
| DATA MANAGEMENT AND STATISTICAL ANALYSIS | Usman Baber, MD MS, Melissa Aquino, MS |
| TRIAL STATISTICIAN | Melissa Aquino, MS |
| TRIAL CHIEF INVESTIGATOR | David E. Kandzari, MD |
| ARO (Academic Research Organization) -Director | Roxana Mehran, MD |
| Angiographic Core Laboratory | Jeffery Popma, MD |
| SAE REPORTING | Theresa Franklin-Bond |
| SAP AUTHOR | Jaya Chandrasekhar, MBBS, MS; Sabato<br>Sorrentino, MD, PhD; Melissa Aquino, MS;<br>Usman Baber, MD, MS |

## SAPPHIRE II PRO



Protocol Number: VP-0714

16 Feb 2017, Clinical Protocol V 1.0

#### Statistical Analysis Plan Signature Page

#### Sapphire II PRO US Clinical Study Protocol Ø1.0mm and 1.25mm Protocol Number: VP-0714

Sponsor: OrbusNeich Medical

Date: September 25, 2017

Version: 1.0

We, the undersigned, have read and approve this Statistical Analysis Plan and agree to its content.

Sponsor Representative

OCOBER 17, 2017
Date

ARO Director, Roxana Mehran, MD

October 13,2017

Date

ARO Biometrics Director, Usman Baber, MD MS

Date

## SAPPHIRE II PRO Protocol Number: VP-0714 16 Feb 2017, Clinical Protocol V 1.0



#### 1. Table of Contents

| 1 | Tal | ole of Contents | 3 |
|---|-----|-----------------------------------------------|---|
| 2 | Ab | breviations and Definitions | 4 |
| 3 | Int | roduction | 5 |
| | 3.1 | Study Investigated Device | 5 |
| | 3.2 | Purpose of the analyses | 5 |
| 4 | Stu | dy Overview (Design/Population/Timeline) | 5 |
| | 4.1 | Selection for Entry into the Study | 6 |
| | 4.2 | Subject Withdrawal Criteria | 6 |
| 5 | End | dpoints | 7 |
| | 5.1 | Primary Endpoint | 7 |
| | 5.2 | Secondary Endpoints | 7 |
| | | 5.2.1 Procedure–Related | 7 |
| | | 5.2.2In-hospital Clinical Safety and Efficacy | 8 |
| 6 | Stu | dy Variables | 9 |
| 7 | An | alysis Populations 1 | 9 |
| | 7.1 | Full Analysis Population | 9 |
| 8 | S | Summary of Study Data2 | 0 |
| | 8.1 | Listing of tables and mock tables | 1 |

## SAPPHIRE II PRO Protocol Number: VP-0714 16 Feb 2017, Clinical Protocol V 1.0



## 2. Abbreviations and Definitions

| ΛE | adverse event |
|------|------------------------------------------------|
| CEC | Clinical Events Committee |
| CRF | case report form |
| FDA | Food and Drug Administration |
| ICF | informed consent form |
| ICH | International Committee of Harmonization |
| IDE | Investigational Device Exemption |
| IRB | Institutional Review Board |
| MI | myocardial infarction |
| PCI | percutaneous coronary intervention |
| PTCA | Percutaneous Transluminal Coronary Angioplasty |
| QCA | quantitative coronary angiography |
| SAE | serious adverse event |
| TIMI | Thrombolysis In Myocardial Infarction |
| TLF | target lesion failure |
| TLR | target lesion revascularization |
| TVF | target vessel failure |
| TVR | target vessel revascularization |
| UADE | unanticipated adverse device event |

## SAPPHIRE II PRO Protocol Number: VP-0714 16 Feb 2017, Clinical Protocol V 1.0



#### 3.Introduction

#### 3.1Study Investigational Device

The Sapphire® II PRO Coronary Dilatation Catheter is a percutaneous transluminal coronary angioplasty (PTCA) balloon catheter with a working length of 140cm. The proximal shaft is a PTFE coated stainless steel hypotube. Hydrophilic lubricious coatings are applied to the distal section. The semi-compliant balloons are made of Nylon 12, available in diameters from 1.0 and 1.25 mm and lengths from 5-15mm, and can be inflated by injecting dilute contrast media solution through the trailing hub of the catheter. The nominal inflation pressure is 6 ATM and the rated burst pressure is 14 ATM. One radiopaque platinum marker band is centrally located within the balloon segment. The catheter is compatible with 5F or larger guiding catheters. The internal lumen of the catheter accepts a standard 0.014 inch PTCA guidewire. The proximal portion of the guidewire enters the catheter tip and advances coaxially out the catheter proximal port, thereby allowing both coaxial guidance and rapid exchange of catheters with a single standard length guidewire. Two marked sections are located on the hypotube shaft to indicate catheter position relative to the tip of either a brachial or femoral guiding catheter. The design of this dilatation catheter does not incorporate a lumen for distal dye injections or distal pressure measurements.

### 3.2.Purpose of the analyses

To assess the acute safety and device procedural success of the 1.0 and 1.25mm diameter Sapphire II PRO dilatation catheter in its intended use for the initial dilatation of coronary artery or by-pass graft stenosis (>70% diameter stenosis).

#### 4.STUDY OVERVIEW

### Study Plan/Design

A prospective, open label, multi-center, single arm, observational study designed to evaluate the acute safety and device procedural success of the Sapphire II PRO Ø1.0 and 1.25 mm PTCA dilatation catheters in subjects with stenotic coronary arteries or bypass grafts during percutaneous coronary intervention.

Statistical Analysis Plan Protocol Number: VP-0714

### SAPPHIRE II PRO 16 Feb 2017, Clinical Protocol V 1.0



#### Study Population, Sites and Timeline.

The target study population is subjects with evidence of ischemia and clinically indicated for one- or two-vessel revascularization procedures by percutaneous coronary intervention.

Sixty (60) subjects will be treated at up to 5 U.S. sites with the Sapphire II PRO  $\emptyset$  1.0 and 1.25 mm PTCA dilatation catheters to pre-dilate coronary arteries or bypass grafts during their index procedure. All subjects will be screened according to the protocol inclusion and exclusion criteria and will be followed through hospital discharge.

#### 4.1. Selection for Entry into the Study

Once the subjects have signed the Institutional Review Board (IRB) approved study informed consent form (ICF) and research authorization forms (RA/HIPAA) and have met all general inclusion and exclusion criteria shown in the protocol, the subjects will be considered eligible to be enrolled in the study to receive treatment with the either the 1.0 or 1.25 mm diameter Sapphire II PRO dilatation catheter. A subject is considered enrolled in the study upon insertion of the investigational device into a guide catheter. Upon enrolment, a subject identification number will be assigned to each subject in a consecutive manner within each clinical site.

#### 4.2. Subject Withdrawal Criteria

Each enrolled subject shall remain in the study until completion of the required follow-up period, however, a subject's participation in any clinical study is voluntary and the patient has the right to withdraw at any time without penalty or loss of benefit. Conceivable reasons for discontinuation may include, but not be limited to, the following:

- Subject death
- Subject voluntary withdrawal
- Subject withdrawal by physician as clinically indicated
- Subject lost-to follow-up

Statistical Analysis Plan Protocol Number: VP-0714

## SAPPHIRE II PRO 16 Feb 2017, Clinical Protocol V 1.0



The reason for subject discontinuation must be documented on the CRF and source documents. The Primary Investigators must also report all subject discontinuations to their IRB, MEC, or HREC as defined by their Institution's procedure.

#### 5.Endpoints

#### 5.1.Primary Endpoint

The study primary end-point shall be defined as Device Procedural Success consisting of a composite of the following parameters:

- · Successful delivery, inflation, deflation and withdrawal of the study balloon
- No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in TIMI flow from baseline related to the study balloon
- Final TIMI flow grade of 3 at the conclusion of the PCI procedure

#### 5.2.Secondary Endpoints

#### 5.2.1.Procedure-Related

The following peri-procedural end-points of study device effectiveness will be determined:

- Successful delivery, inflation, deflation, and withdrawal of the study balloon
- Absence of vessel perforation, flow limiting dissection (grade C or higher, or reduction in TIMI flow from baseline related to the study balloon
- Absence of balloon rupture of the study balloon
- Improvement in Minimum Lumen Diameter (MLD) following pre-dilatation with Sapphire II PRO Ø 1.0 and 1.25 mm PTCA dilatation catheters (measured by QCA)
- And Lesion Success defined as successful PCI in the absence of vessel perforation, flow limiting dissection (grade C or higher, reduction in TIMI flow from baseline related to the study balloon, or clinically significant arrhythmias

#### 5.2.2.In-hospital Clinical Safety and Efficacy

The following end-points will be measured through hospital discharge:

In-hospital Major Adverse Cardiac Events (MACE), a composite of:

## SAPPHIRE II PRO



Protocol Number: VP-0714

16 Feb 2017, Clinical Protocol V 1.0

- All death (cardiac and non-cardiac)
- o Myocardial infarction (MI)
- Target Lesion Revascularization (TLR), clinically indicated
- Individual components of the MACE composite end-point
- In-hospital Target Lesion Failure (TLF) a composite of:
  - o Cardiac death
  - Target vessel MI
  - o TLR, clinically indicated
- In-hospital stent thrombosis (ST) within the target vessel
- Clinically significant arrhythmias (requiring intervention)

## SAPPHIRE II PRO Protocol Number: VP-0714 16 Feb 2017, Clinical Protocol V 1.0



## 6.Study Variables

The SAPPHIRE II PRO study variables consist of information blocks containing baseline data, information about the procedure, and clinical events up to discharge. Statistical Analysis Plan
Protocol Number: VP-0714

## SAPPHIRE II PRO 16 Feb 2017, Clinical Protocol V 1.0



### 7. Analysis Populations

#### 7.1. Full Analysis Population

This study is designed as a single-arm observational trial. The study sample size is based upon treatment of a reasonable number of subjects with the study device to provide a reliable and meaningful assessment of device performance, rather than based upon any statistical hypothesis of an endpoint.

All analyses will be performed on an intent-to-treat basis. The baseline demographic and lesion characteristics and angiographic and clinical outcomes will be evaluated by descriptive statistics. These calculations will be performed under the assumption that the data are in a normal distribution. All enrolled subjects will be analyzed on an intent-to-treat (ITT) basis as well as per protocol criteria.

#### 7.2 Summary of Study Data

The baseline demographic and lesion characteristics and angiographic and clinical outcomes will be evaluated by descriptive statistics. These calculations will be performed under the assumption that the data are in a normal distribution. All continuous variables will be summarised using the following descriptive statistics: n (non-missing sample size), mean and standard deviation. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. Deaths, Serious Adverse Events and other Significant Adverse Events will be reported as number and percentage. All analyses will be performed using SAS version 9.4 (NC, USA).

Lesion related outcomes were assessed using core lab data. Where core lab was not analyzable, site reported data were used. No outcomes were imputed.

## 8.1. Listing of Tables and mock tables

This section gives details on mock tables.

Table Listings

| Number | Table Title | Summary Statistics |
|---|---|---|
| 1 | Primary end-point | n (%) |
| 2 | Secondary end-points | n (%) |
| 3 | Summary of baseline patient characteristics | n, mean, SD, Median, min,<br>max,<br>n (%) |
| 4 | Summary of discharge patient data | n, mean, SD, Median, min,<br>max,<br>n (%) |
| 5 | Summary of procedural patient characteristics | n, mean, SD, Median, min,<br>max,<br>n (%) |
| 6 | Summary of site reported lesion level Data | n, mean, SD, Median, min,<br>max,<br>n (%) |
| 7 | Core lab lesion level data | n, mean, SD, Median, min,<br>max,<br>n (%) |
| 8 | Lesion level study outcomes | n, mean, SD, Median, min,<br>max,<br>n (%) |
| 9 | In-hospital patient level outcomes | n (%) |

Table 1: Primary End-Point:

| | Overall population N = patients |
|---|---|
| Primary Endpoint | |
| Successful balloon delivery to the target lesion | |
| No | |
| Yes | |
| Successful inflation at the target lesion | |
| No | |
| Yes | |
| Successful deflation and withdrawal of the study balloon | |
| No | |
| Yes | |
| Vessel Perforation | |
| No | |
| Yes | |
| Flow limiting dissection (Grade C or Higher) | |
| No | |
| Yes | |
| No reduction in TIMI flow from baseline related to the study balloon (i.e. TIMI>=0) | |
| No | |
| Yes | |
| Final TIMI flow grade of 3 at the conclusion of the PCI procedure | |
| No | |
| Yes | |

Table 2: Secondary End-Points:

| | Overall population N = patients |
|---|---|
| Successful balloon delivery to the target lesion | |
| No | |
| Yes | |
| Successful inflation at the target lesion | |
| No | |
| Yes | |
| Successful deflation and withdrawal of the study balloon | |
| No | |
| Yes | |
| Vessel Perforation | |
| No | |
| Yes | |
| Flow limiting dissection (Grade C or Higher) | |
| No | |
| Yes | |
| No reduction in TIMI flow from baseline related to the study balloon (i.e. TIMI>=0) | |
| No | |
| Yes | |
| Final TIMI flow grade of 3 at the conclusion of the PCI procedure | |
| No | |
| Yes | |
| Balloon rupture of the study balloon | |
| No | |
| Yes | |
| Improvement in Minimum Lumen Diameter | |
| No | |
| Yes | |
| Lesion success | |
| No | |
| Yes | |
| Vessel Perforation | |
| No | |
| Flow limiting dissection (Grade C or Higher) | |
| No | |
| Yes | |
| No reduction in TIMI flow from baseline related to the study balloon (i.e. TIMI>=0) | |
| No | |
| Yes | |

| | Overall population N = patients |
|----------------------------------|---------------------------------|
| Clinically Significant Arrythmia | |
| No | |
| Yes | |

Table 3: Baseline patient characteristics:

| | Overall population N = patients |
|---|---|
| CLINICAL CHARACTERISTICS | pationto |
| Age (Years) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | ****** |
| Median (IQR) | |
| Gender | |
| Female | - In- The |
| Male | |
| Race | |
| Asian | |
| Black | |
| White | |
| BMI (kg/m²) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Diabetes Mellitus | |
| No No | |
| Yes | |
| Diabetes Treatment | |
| Diet | |
| Insulin | |
| None | |
| Oral Medication | |
| Current Cigarette smoking (within 30 days) | |
| No | |
| Yes | |
| Hypercholesterolemia (requiring treatment) | |
| -No | |
| Yes | |
| Hypertension (requiring treatment) | |
| No I | |
| Yes | |
| Peripheral arterial disease (arms, legs, renal, mesenteric, aneurysm) | |
| No | |
| Yes | |
| Previous history of stroke more than 6 months prior | |

| | Overall<br>population<br>N =<br>patients |
|---|---|
| No | |
| Yes | |
| Prior myocardial infarction | |
| No | |
| Yes | |
| Previous PCI | |
| No | |
| Yes | |
| Previous CABG | |
| No | |
| Yes | |
| Left ventricular ejection fraction | |
| 30-40% | |
| >40% | |
| Unknown | |
| Angina status | |
| Asymptomatic | |
| NSTEMI | |
| Stable angina | |
| Unstable angina | |
| CCS Class | |
| 0 | |
| 1 | |
| II | |
| III | |
| IV | |
| Heart failure NYHA class III or IV | |
| No | |
| Yes | |
| Extent of coronary artery disease (number of vessels with CAD >= 50%) | |
| 1 | |
| 2- | |
| 3 | |
| BASELINE MEDICATIONS | |
| ACE inhibitors or ARB | |
| No | |
| Yes | |
| Beta-blockers | |
| No | |
| Yes | |
| Calcium channel blockers | |

| | Overall population N = patients |
|---------------------------------------|---------------------------------|
| No | |
| Yes | |
| Long-acting nitrate | |
| No | |
| Yes | |
| Ranexa | |
| No | |
| Yes | |
| Oral Anticoagulation | |
| No | |
| Yes | |
| Statins | |
| No | |
| Yes | |
| Proton pump inhibitor | |
| No | |
| Yes | |
| Aspirin | |
| No | |
| Yes | |
| P2Y12 inhibitor | |
| Clopidogrel | |
| None | |
| Prasugrel | |
| Ticagrelor | |
| BASELINE LABS | |
| Creatinine | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Hemoglobin | F |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| White cell count (10 <sup>9</sup> /L) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |

| | Overall population N = patients |
|-------------------------------------|---------------------------------|
| Platelets | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Troponin | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| СКМВ | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| BASELINE ECG | |
| 12-lead electrocardiogram performed | |
| No | |
| Yes | |
| Rhythm | |
| AF/flutter | |
| Other | |
| Sinus Rhythm | |
| Q wave | |
| No | |
| Yes -Existing | |
| ST-segment depression or elevation | |
| No | |
| Yes - Existing | |
| Yes - New | |

Table 4: Discharge patient data

| | Overall<br>population<br>N =<br>patients |
|---|---|
| DISCHARGE | |
| Did any complications occur before discharge | |
| No | |
| Did the patient complete all study related activities at the time of discharge? | |
| No | |
| Yes | |
| Was there a protocol deviation? | |
| No | |
| Yes | |
| DISCHARGE CARDIAC ENZYMES | |
| Troponin | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| CKMB (Immediately after procedure) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| CKMB (6-12h after PCI) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| CKMB (18-24h after PCI or prior to discharge) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| POST PCI LABS | |
| Lowest Hemoglobin value | |
| N, N Missing | |
| Mean ± Std | an e-metric |
| Min , Max | |
| Median (IQR) | |
| Highest Creatinine value | |
| N, N Missing | |
| Mean ± Std | |

| | Overall population N = patients |
|--------------------------------------------|---------------------------------|
| Min , Max | |
| Median (IQR) | |
| Patient required new hemodialysis post-PCI | |
| Missing | |
| No | |
| POST PCI ECG | |
| 12-lead electrocardiogram performed | |
| No | |
| Yes | |
| Rhythm | |
| AF/flutter | |
| Other | |
| Sinus Rhythm | |
| Q wave | |
| No | |
| Yes - Existing | |
| ST-segment depression or elevation | |
| No | |
| Yes - Existing | |
| POST PCI MEDICATIONS | |
| ACE inhibitors or ARB | |
| No | |
| Yes | |
| Beta-blockers | |
| No | |
| Yes | |
| Calcium channel blockers | |
| No | |
| Yes | |
| Long-acting nitrate | |
| No | |
| Yes | |
| Ranexa | |
| No | |
| Yes | |
| Oral Anticoagulation | |
| No | |
| Yes | |
| Statins | |
| No | |
| Yes | |

| 25 | Overall population N = patients |
|-----------------------|---------------------------------|
| Proton pump inhibitor | |
| No | |
| Yes | |
| Aspirin | |
| No | |
| Yes | |
| P2Y12 inhibitor | |
| Clopidogrel | |
| None | |
| Prasugrel | |
| Ticagrelor | |

Table 5: Procedural patient characteristics

| | Overall population N = patients |
|---|---|
| PROCEDURAL CHARACTERISTICS | |
| Number of lesions per patients | |
| Multiple | |
| Single | |
| Extent of coronary artery disease (number of vessels with CAD >= 50%) | |
| 1 | |
| 2 | |
| 3 | |
| Presence of Left main disease >= 50% | |
| No | |
| Yes | |
| Total contrast volume used (diagnostic and intervention) (ml) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Procedure duration (min) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Total fluroscopy time (min) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Specify arterial sheath access | |
| Femoral | |
| Radial | |
| Procedural medication (within 72 hours of PCI) | |
| Bivalirudin | |
| Low molecular weight heparin | |
| Unfractionated heparin | |
| Heart rate(beats per min) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |

#### VP-0714

| | Overall population N = patients |
|--------------------------------|---------------------------------|
| Systolic Blood Pressure(mmHg) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Diastolic Blood Pressure(mmHg) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |

Table 6: Lesion level data (Site reported)

| | Overall population N = lesions |
|---|---|
| LESION CHARACTERISTICS | |
| SAPPHIRE II PRO Device size | |
| 1.0 x 10 mm | |
| 1.0 x 15 mm | |
| 1.0 x 8 mm | |
| 1.25 x 10 mm | |
| 1.25 x 15 mm | |
| 1.25 x 5 mm | |
| 1.25 x 8 mm | |
| Vessel treated | |
| Bypass graft | |
| Diagonal branch of LAD | |
| LAD | 1102 - N. 1 - 1 |
| LCx | |
| Marginal branch of LCx | |
| Posterior descending branch of RCA | |
| RCA | |
| Lesion location | 3, |
| Distal | |
| Mid | |
| Ostial | |
| Prox | |
| Number of inflations per lesion | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| Successful baloon delivery to the target lesion | |
| Yes | |
| Successful baloon inflation and deflation at the target lesion | |
| No | |
| Yes | |
| Inflation pressure (atm) | 1 |
| N, N Missing | |
| Mean ± Std | 19 1 150 |
| Min , Max | |
| Median (IQR) | |
| Number of inflations per lesion | |
| 01 | |

| | Overall population N = lesions |
|---|---|
| 02 | |
| 03 | |
| 04 | |
| 05 | |
| 06 | |
| Was there balloon rupture? | |
| No | |
| Yes | |
| Successful withdrawal of the balloon from the target lesion | |
| Yes | |
| Was any post-dilation performed with stent implantation? | |
| No | |
| Not applicable | |
| Yes | |
| Was post procedural TIMI flow <3 at any lesion? | |
| No | |
| Yes | |
| Stent type implanted | |
| Biodegradable polymer stent (eg. Synergy) | |
| None | |
| Other | |
| Resolute | |
| Xience | |
| Stent implanted | |
| No | |
| Yes | |

Table 7: Core lab lesion level data

| | Overall<br>population<br>N =<br>lesions |
|--------------------------|-----------------------------------------|
| CASS Segment | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| CORE LAB | |
| Lesion location | |
| Missing | |
| Distal | |
| Mid | |
| Ostial | |
| Prox | |
| Lesion Length analyzable | |
| Missing | |
| No | |
| Lesion length (mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Eccentricity | |
| Missing | |
| Concentric | |
| Eccentric | |
| Thrombus | |
| Missing | |
| No | |
| Yes | |
| Tortuosity | |
| Missing | |
| None | |
| Calcification | |
| Missing | |
| Mod | |
| None | |
| Not-analyzable | |
| Severe | |
| Ulceration | |
| Missing | |

. .

| | Overall population N = lesions |
|-------------------------------------|--------------------------------|
| No | |
| Yes | |
| Aneurysm | |
| Missing | |
| No | |
| Intimal Flap | |
| Missing | |
| No | |
| Pre TIMI | |
| Missing | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| Number of frames | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Bifurcation | |
| Missing | |
| No | |
| Yes | |
| Prox Main branch | |
| Missing | |
| No | |
| Not-analyzable | |
| Yes | |
| Distal Main branch | |
| Missing | |
| No | |
| Not-analyzable | |
| Yes | |
| Side branch | |
| Missing | |
| No | |
| Not-analyzable | |
| Yes | |
| Branch diameter stenosis analyzable | |
| Missing | |
| No | |

| | Overall population N = lesions |
|-----------------------------|--------------------------------|
| Yes | |
| Branch diameter stenosis, % | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Prox Normal analyzable | |
| Missing | |
| No | |
| Prox Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Distal Normal analyzable | |
| Missing | |
| No | |
| Distal Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| MLD analyzable | |
| Missing | |
| No | |
| MLD(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Prox Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Prox Normal(mm) | |
| N, N MissIng | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Distal Normal analyzable | |
| Missing | |

| | Overall population N = lesions |
|------------------------------|-----------------------------------------|
| No | |
| Yes | |
| Distal Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| MLD analyzable | |
| Missing | |
| No | |
| Yes | |
| MLD(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| CORONARY DILATATION CATHETER | |
| Aneurysm | |
| MissIng | |
| No | |
| Not-analyzable | |
| Post TIMI | |
| 1 | |
| 2 | |
| 3 | |
| Number of frames analyzable | |
| Missing | |
| No | |
| Yes | |
| Number of frames | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | 1997-1997-1997-1997-1997-1997-1997-1997 |
| Median (IQR) | |
| No Reflow | |
| Missing | |
| No . | |
| Not-analyzable | |
| Abrupt closure | |
| Missing | |
| No | |

| | Overall<br>population<br>N =<br>lesions |
|------------------------------|------------------------------------------|
| Not-analyzable | |
| Dissection | |
| 0 | |
| Stalning | |
| Missing | |
| Not-analyzable | |
| Dissection Length analyzable | |
| Missing | |
| No | |
| Dissection Length (mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | THE SAME AND SAME AND |
| Median (IQR) | 77-2- |
| Branch % stenosis analyzable | |
| Missing | |
| No | |
| Yes | |
| Branch % Stenosis | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Distal embolus | |
| Missing | |
| No | |
| Not-analyzable | |
| Perforation | |
| No | |
| Spasm | |
| Missing | |
| No | |
| Not-analyzable | 10-10-10-10-10-10-10-10-10-10-10-10-10-1 |
| PROJECTION #1 | |
| Prox Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Prox Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |

| | Overall<br>population<br>N =<br>lesions |
|--------------------------|-----------------------------------------|
| Min , Max | |
| Median (IQR) | |
| Distal Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Distal Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| MLD analyzable | |
| Missing | |
| No | |
| Yes | |
| MLD(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| PROJECTION #2 | |
| Prox Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Prox Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | 52<br>52 |
| Distal Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Distal Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| MLD analyzable | |
| Missing | |

| | Overall population N = lesions |
|-----------------------------|--------------------------------|
| No | |
| Yes | |
| MLD(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| FINAL POST-PROCEDURE | |
| Thrombus | |
| Missing | |
| No | |
| Not-analyzable | |
| Aneurysm | |
| Missing | |
| No | |
| Not-analyzable | |
| Post TIMI | |
| 0 | |
| 3 | |
| Number of frames analyzable | |
| Missing | |
| No | |
| Yes | |
| Number of frames | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| No Reflow | |
| Missing | |
| No | |
| Abrupt closure | |
| Missing | |
| No | |
| Yes | |
| Dissection | |
| Missing | |
| 0 | |
| Staining | |
| Missing | |
| Not-analyzable | |

| | Overall<br>population<br>N =<br>lesions |
|------------------------------|-----------------------------------------|
| Dissection Length analyzable | |
| Missing | |
| Yes | |
| Dissection Length(mm) | |
| Missing | |
| Branch % stenosis analyzable | |
| Missing | |
| No | |
| Yes | |
| Distal embolus | |
| Missing | |
| Yes | |
| Perforation | |
| Missing | |
| No | |
| Spasm | |
| Missing | |
| No | |
| PROJECTION #1 | |
| Prox Normal analyzable | |
| Missing | * |
| No | |
| Prox Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Distal Normal analyzable | |
| Missing | |
| No | |
| Distal Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| MLD analyzable | |
| Missing | |
| No | |
| MLD(mm) | |
| N, N Missing | |
| Mean ± Std | |

| | Overall population N = lesions |
|--------------------------|--------------------------------|
| Min , Max | |
| Median (IQR) | |
| PROJECTION #2 | |
| Prox Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Prox Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Distal Normal analyzable | |
| Missing | |
| No | |
| Yes | |
| Distal Normal(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| MLD analyzable | |
| Missing | |
| No | |
| Yes | |
| MLD(mm) | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |

Table 8: Lesion level study outcomes

| | Overall population N = lesions |
|---|---|
| Device related primary endpoint composite | |
| Successful delivery, inflation, deflation and withdrawal of the study balloon | |
| No | |
| Yes | |
| Successful delivery | |
| No | |
| Yes | |
| Inflation | |
| No | |
| Yes | |
| Withdrawal of the study balloon | |
| No | |
| Yes | |
| No evidence of vessel perforation, flow limiting dissection (grade C or higher) or reduction in TIMI | |
| No | |
| Yes | |
| Vessel perforation | |
| No | |
| Yes | |
| Lesion Success | |
| No | 7 |
| Yes | |
| Vessel perforation | |
| No | |
| Yes | |
| Flow limiting dissection (grade C or higher) | |
| No | |
| Yes | |
| Flow limiting dissection (grade C or higher) | |
| No | |
| Yes | |
| Clinically significant arrhythmia | |
| No | |
| Yes | |
| No reduction in TIMI flow from baseline related to the study balloon (i.e. TIMI>=0) | |
| No | |
| Yes | |
| No reduction in TIMI flow from baseline related to the study balloon (i.e. TIMI>=0) | |
| No | |

| | Overall population N = lesions |
|---|---|
| Yes | |
| Change in Minimum lumen diameter, pre and post balloon dilation | |
| N, N Missing | |
| Mean ± Std | |
| Min , Max | |
| Median (IQR) | |
| Final TIMI flow grade of 3 at the conclusion of the PCI procedure | |
| No | |
| Yes | |
| Improvement in Minimum Lumen Diameter | |
| No | |
| Yes | |
| Balloon rupture | |
| No | |
| Yes | |

Table 9: In-hospital patient level outcomes

| | Overall population N = patients |
|---|---|
| MACE, composite of all death, MI or clinically indicated TLR | |
| Death | |
| MI | |
| Clinically indicated TLR | |
| Target lesion failure, composite of cardiac death, target vessel MI or clinically indicated TLR | |
| Stent thrombosis within the target vessel | |
| Clinically significant arrhythmias requiring intervention | |
| Device related Primary composite endpoint | |